CLINICAL TRIAL: NCT00303914
Title: A Survey of Disease and Treatment-Related Symptoms in Patients With Invasive Cancer: Prevalence, Severity and Treatment
Brief Title: Study of Symptoms Caused by Cancer and Cancer Therapy in Patients With Invasive Breast, Lung, Prostate, or Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000462104; ECOG-E2Z02
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer; Cognitive/Functional Effects; Colorectal Cancer; Lung Cancer; Pain; Prostate Cancer; Psychosocial Effects of Cancer and Its Treatment
Keywords: pain; psychosocial effects of cancer and its treatment; cognitive/functional effects; recurrent breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent colon cancer; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; recurrent rectal cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer; extensive stage small cell lung cancer; limited stage small cell lung cancer; recurrent small cell lung cancer; recurrent non-small cell lung cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent prostate cancer; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer; male breast cancer; pulmonary carcinoid tumor
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Pain; Prostatic Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms, Male | interventions — Mental Status and Dementia Tests; Psychiatric Rehabilitation

INTERVENTIONS:
Procedure: assessment of therapy complications
Procedure: cognitive assessment
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: Questionnaires that assess symptoms caused by cancer and cancer therapy may help improve the ability to plan treatment for patients with invasive cancer to help them live longer and more comfortably.

PURPOSE: This clinical trial is studying symptoms caused by cancer and cancer therapy in patients with invasive breast, lung, prostate, or colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the prevalence, severity, and interference due to physical and psychological symptoms experienced (over a 4 to 5 week period) by patients with invasive primary breast, lung, prostate, or colorectal cancer who are being followed on an outpatient basis at ECOG institutions.

Secondary

* Determine if the number of symptom-related interventions are related to the providers' perception of symptom severity.
* Determine whether physical symptoms are more commonly prioritized and treated compared to psychological symptoms.
* Determine the percentage of patients who experience a significant reduction in moderate-to-severe symptoms and characterize the determinants of symptom relief.
* Determine the focus and scope of interventions chosen by oncologists to improve the symptom control of patients seen in outpatient clinics.

OUTLINE: This is an open-label, multicenter study. Patients are stratified according to disease type, prevalence according to gender, race/ethnicity, age, and type of treatment.

Patients complete the M.D. Anderson Symptom Assessment Inventory and other questionnaires, rating the symptoms most frequently found in this patient group and how much these symptoms interfere with mood and activity-related domains, on day 1 and again between days 28-35.

At the same time points, a healthcare provider (treating physician, nurse, or physician assistant) completes the Revised Edmonton Staging System for Cancer Pain questionnaire, assessing the patient's cancer pain on the basis of mechanism of pain, incidental pain, psychological distress and addictive behavior, and cognitive function, for clinical prognosis on pain control.

PROJECTED ACCRUAL: A total of 2,310 patients and their physicians will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Being seen in an outpatient setting at an ECOG-affiliated academic institution, a CGOP site, or a CCOP site

  * In pretreatment, active treatment, or follow-up for their cancer
* Clinically diagnosed invasive cancer involving at least 1 of the following primary sites:

  * Breast
  * Lung
  * Prostate
  * Colorectal
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Male or female
* Menopausal status not specified
* Willing to complete a written survey between day 28 and day 35 after completion of the baseline assessment
* Able to read, write, and understand English
* No significantly impaired cognitive status which, in the opinion of the investigator, would hinder ability to provide responses

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2310 (Estimated)
Dates: Start 2006-03-14 (Actual); Primary Completion 2008-03 (Actual); Study Completion 2013-03-04 (Actual)

PRIMARY OUTCOMES:
Prevalence, severity, and interference due to physical and psychological symptoms experienced by cancer patients as assessed by MD Anderson Symptom Inventory at baseline and days 28-35 following initial assessment

SECONDARY OUTCOMES:
Number of symptom-related interventions related to the providers perception of symptom severity as assessed by The Revised Edmonton Staging System for cancer pain (rESS) at baseline and days 28-35 following initial assessment
Compare treatment priority based on physical or psychological symptoms
Percentage of patients who experience a significant reduction in moderate-to-severe symptoms and characterize the determinants of symptom relief
Focus and scope of interventions chosen to improve symptom control

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Fisch, MD, MPH, FACP, Study Chair — M.D. Anderson Cancer Center; Charles Cleeland, PhD — M.D. Anderson Cancer Center
Locations (32):
- United States (32):
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Evanston Hospital, Evanston, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota

REFERENCES:
- [Result] Manola J, Zhao F, Miller AH, et al.: Patterns of antidepressant use in cancer patients (pts): An analysis from SOAPP (ECOG E2Z02: Symptom Outcomes and Practice Patterns). [Abstract] J Clin Oncol 30 (Suppl 15): A-9016, 2012.
- [Result] Zhao F, Wagner LI, Pirl WF, et al.: Racial disparities in depressive symptom prevalence and selective serotonin reuptake inhibitor (SSRI) utilization in cancer patients: An analysis from ECOG E2Z02: Symptom Outcomes and Practice Patterns (SOAPP). [Abstract] J Clin Oncol 30 (Suppl 15): A-6076, 2012.
- [Result] Wagner LI, Zickl L, Smith ML, et al.: Prospective assessment of symptom burden among cancer survivors with common solid tumors: results from ECOG trial E2Z02. [Abstract] J Clin Oncol 29 (Suppl 15): A-9137, 2011.
- [Result] Hamann HA, Lee J, Schiller JH, et al.: Clinician perceptions of care difficulty and quality of life for lung cancer patients: results from the ECOG SOAPP study (E2Z02). [Abstract] J Clin Oncol 28 (Suppl 15): A-9102, 2010.
- [Result] Tevaarwerk A, Lee J, Sesto MC, et al.: Predictors of employment (empl) outcomes in outpatients (pts) with common solid tumors: A secondary analysis from E2Z02 (ECOG's SOAPP study). [Abstract] J Clin Oncol 28 (Suppl 15): A-9118, 2010.
- [Derived] Zhao F, Chang VT, Cleeland C, Cleary JF, Mitchell EP, Wagner LI, Fisch MJ. Determinants of pain severity changes in ambulatory patients with cancer: an analysis from Eastern Cooperative Oncology Group trial E2Z02. J Clin Oncol. 2014 Feb 1;32(4):312-9. doi: 10.1200/JCO.2013.50.6071. Epub 2013 Dec 23. PMID 24366929